CLINICAL TRIAL: NCT02135952
Title: Metronidazole and Amoxicillin as Adjuncts to Scaling and Root Planing for the Treatment of Type 2 Diabetic Subjects With Periodontitis: a Randomized Placebo-controlled Clinical Trial
Brief Title: Metronidazole and Amoxicillin for the Treatment of Type 2 Diabetic Subjects With Periodontitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Guarulhos (Other)
Responsible Party: Principal Investigator, Poliana Mendes Duarte, PhD, University of Guarulhos
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SISNEP/697; 2013/01072-5 (Other Grant/Funding Number: FAPESP - 2013/01072-5)
Record Dates: First submitted 2014-05-05; First posted 2014-05-12 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Periodontitis
Keywords: Periodontitis; Diabetes
MeSH Terms: conditions — Periodontitis; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SRP+MTZ+AMX (Active Comparator): Scaling and root planing (SRP) + metronidazole (MTZ; 400 mg thrice a day [TID] for 14 days) + amoxicillin (AMX; 500 mg TID for 14 days)
  Interventions: Procedure: SRP; Drug: MTZ+AMX
- SRP+placebo (Placebo Comparator): Scaling and root planing + placebo
  Interventions: Procedure: SRP; Other: Placebo

INTERVENTIONS:
Procedure: SRP — SRP in four to six appointments lasting approximately 1 h each, using manual curettes and ultrasonic device under local anesthesia.
Other: Placebo — Administration of placebo for 14 days started immediately after the first session of SRP.
  Arms: SRP+placebo
Drug: MTZ+AMX — Administration of antibiotics (metronidazole and amoxicillin) for 14 days started immediately after the first session of SRP.
  Arms: SRP+MTZ+AMX

SUMMARY:
Diabetes mellitus (DM) is a widely prevalent disease associated with several major systemic and oral complications, such as periodontitis. The use of adjunctive local and/or systemic antimicrobials has been proposed to improve the clinical and glycemic outcomes of the scaling and root planing (SRP) in diabetic subjects. The combination of metronidazole (MTZ) and amoxicillin (AMX) has been largely recognized as an effective therapy for improving the clinical and microbiological outcomes of SRP in the treatment of with chronic periodontitis (ChP). However, no previous clinical trials to date have evaluated the effects of this antibiotic combination in the treatment of diabetic subjects with periodontitis. Therefore, the aim of this randomized clinical trial (RCT) will be to evaluate the clinical and microbiological effects of the use of MTZ+AMX as adjuncts to SRP for the treatment of type 2 diabetic subjects with generalized ChP.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 35 years of age
* Diagnosis of type 2 DM for ≥ 5 years
* DM treatment with diet and insulin supplementation or oral hypoglycemic agents
* Glycated hemoglobin (HbA1c) levels ≥ 6.5% ≤ 11%
* At least 15 teeth
* More than 30% of the sites with probing depth (PD) and clinical attachment level (CAL) ≥ 4 mm
* Minimum of six teeth with at least one site with PD and CAL ≥ 5 mm and bleeding on probing (BoP) at baseline.

Exclusion Criteria:

* Pregnancy
* Lactation
* Current smoking
* Smoking within the past 5 years
* Scaling and root planing (SRP) in the previous 12 months
* Antimicrobial therapies during the previous 6 months
* Medical conditions requiring prophylactic antibiotic coverage
* Continuous use of mouthrinses containing antimicrobials in the preceding 3 months
* Systemic conditions (except DM) that could affect the progression of periodontitis (e.g. immunological disorders, osteoporosis)
* Long-term administration of anti-inflammatory
* Long-term administration of immunosuppressive medications
* Allergy to metronidazole and/or amoxicillin
* Presence of periapical pathology
* Use of orthodontic appliances
* Presence of extensive prosthetic rehabilitation
* Major complications of DM (i.e. cardiovascular and peripheral vascular diseases [ulcers, gangrene and amputation], neuropathy and nephropathy)

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2011-09; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Changes in number of sites with probing depth (PD) ≥5 mm post-treatment | From baseline to 12 months

SECONDARY OUTCOMES:
PD and clinical attachment level (CAL) changes at initially moderate sites | From baseline to 12 months and from baseline to 24 months
PD and CAL changes at initially deep sites | From baseline to 12 months and from baseline to 24 months
Changes in number of sites with PD ≥5mm | From baseline to 12 months and from baseline to 24 months
Full-mouth PD and CAL | Baseline, 3, 6, 12 and 24 months
Full-mouth percentages of sites with plaque | Baseline, 3, 6, 12 and 24 months
Full-mouth percentages of sites with marginal bleeding | Baseline, 3, 6, 12 and 24 months
Full-mouth percentages of sites with bleeding on probing | Baseline, 3, 6, 12 and 24 months
Full-mouth percentages of sites with suppuration | Baseline, 3, 6, 12 and 24 months
Full-mouth percentages of sites with PD ≥5mm | Baseline, 3, 6,12 and 24 months
Serum levels of glycated hemoglobin (HbA1c) | Baseline, 3, 6, 12 and 24 months
Serum levels of fasting plasma glucose FPG | Baseline, 3, 6, 12 and 24 months
Levels of periodontal pathogenic bacterial species | Baseline, 3, 6, 12 and 24 months
Occurrence of adverse events | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Poliana M Duarte, PhG, Principal Investigator — University of Guarulhos
Locations (1):
- University of Guarulhos, Guarulhos, São Paulo, Brazil

REFERENCES:
- [Background] Amid R, Tabeie MB, Kadkhodazadeh M, Mehdizadeh AR, Youssefi N. Local concentration of systemic amoxicillin and metronidazole in healthy and inflamed gingiva: a comparative in vivo study. Drug Metabol Drug Interact. 2012 May 10;27(2):113-8. doi: 10.1515/dmdi-2012-0003. PMID 22706234
- [Background] Borgnakke WS, Ylostalo PV, Taylor GW, Genco RJ. Effect of periodontal disease on diabetes: systematic review of epidemiologic observational evidence. J Clin Periodontol. 2013 Apr;40 Suppl 14:S135-52. doi: 10.1111/jcpe.12080. PMID 23627324
- [Background] Cionca N, Giannopoulou C, Ugolotti G, Mombelli A. Amoxicillin and metronidazole as an adjunct to full-mouth scaling and root planing of chronic periodontitis. J Periodontol. 2009 Mar;80(3):364-71. doi: 10.1902/jop.2009.080540. PMID 19254119
- [Background] Cionca N, Giannopoulou C, Ugolotti G, Mombelli A. Microbiologic testing and outcomes of full-mouth scaling and root planing with or without amoxicillin/metronidazole in chronic periodontitis. J Periodontol. 2010 Jan;81(1):15-23. doi: 10.1902/jop.2009.090390. PMID 20059413
- [Background] Feres M. Antibiotics in the treatment of periodontal diseases: microbiological basis and clinical applications. Ann R Australas Coll Dent Surg. 2008 Jun;19:37-44. PMID 19728628
- [Background] Feres M, Soares GM, Mendes JA, Silva MP, Faveri M, Teles R, Socransky SS, Figueiredo LC. Metronidazole alone or with amoxicillin as adjuncts to non-surgical treatment of chronic periodontitis: a 1-year double-blinded, placebo-controlled, randomized clinical trial. J Clin Periodontol. 2012 Dec;39(12):1149-58. doi: 10.1111/jcpe.12004. Epub 2012 Sep 27. PMID 23016867
- [Background] Grossi SG, Skrepcinski FB, DeCaro T, Robertson DC, Ho AW, Dunford RG, Genco RJ. Treatment of periodontal disease in diabetics reduces glycated hemoglobin. J Periodontol. 1997 Aug;68(8):713-9. doi: 10.1902/jop.1997.68.8.713. PMID 9287060
- [Background] Jimenez M, Hu FB, Marino M, Li Y, Joshipura KJ. Type 2 diabetes mellitus and 20 year incidence of periodontitis and tooth loss. Diabetes Res Clin Pract. 2012 Dec;98(3):494-500. doi: 10.1016/j.diabres.2012.09.039. Epub 2012 Oct 3. PMID 23040240
- [Background] Lang NP, Tonetti MS. Periodontal risk assessment (PRA) for patients in supportive periodontal therapy (SPT). Oral Health Prev Dent. 2003;1(1):7-16. PMID 15643744
- [Background] Silva MP, Feres M, Sirotto TA, Soares GM, Mendes JA, Faveri M, Figueiredo LC. Clinical and microbiological benefits of metronidazole alone or with amoxicillin as adjuncts in the treatment of chronic periodontitis: a randomized placebo-controlled clinical trial. J Clin Periodontol. 2011 Sep;38(9):828-37. doi: 10.1111/j.1600-051X.2011.01763.x. Epub 2011 Jul 15. PMID 21762197
- [Background] Zandbergen D, Slot DE, Cobb CM, Van der Weijden FA. The clinical effect of scaling and root planing and the concomitant administration of systemic amoxicillin and metronidazole: a systematic review. J Periodontol. 2013 Mar;84(3):332-51. doi: 10.1902/jop.2012.120040. Epub 2012 May 21. PMID 22612369
- [Derived] Tamashiro NS, Duarte PM, Miranda TS, Maciel SS, Figueiredo LC, Faveri M, Feres M. Amoxicillin Plus Metronidazole Therapy for Patients with Periodontitis and Type 2 Diabetes: A 2-year Randomized Controlled Trial. J Dent Res. 2016 Jul;95(7):829-36. doi: 10.1177/0022034516639274. Epub 2016 Mar 24. PMID 27013640